CLINICAL TRIAL: NCT00490503
Title: Non-Invasive MRI and MRS Techniques for Assessing Therapeutic Response to Pre-surgical Chemotherapy in Breast Cancer Patients
Brief Title: Non-Invasive Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy Techniques (MRS) for Assessing Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0501; P50CA116199 (NIH)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; DCE-MRI; DW-MRI; MRS; MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The tissues removed during surgery (mastectomy) will be collected as part of this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI + MRS: Patients with newly diagnosed stage II A-B or III A-C breast cancers who are scheduled to start systemic chemotherapy.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Magnetic Resonance Spectroscopy (MRS)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — 3 Scans performed before chemotherapy, 21 days (plus or minus 3 days) after start chemotherapy (Day 1 = your first day of chemotherapy), and at end of chemotherapy/before surgery.
  Other Names: MRI
Procedure: Magnetic Resonance Spectroscopy (MRS) — 3 MRI Scans with MRS performed before chemotherapy, 21 days (plus or minus 3 days) after start chemotherapy (Day 1 = your first day of chemotherapy), and at end of chemotherapy/before surgery.
  Other Names: MRS

SUMMARY:
The goal of this clinical research study is to learn if magnetic resonance imaging (MRI) with magnetic resonance spectroscopy (MRS) can show the effects of pre-surgical chemotherapy in breast cancer patients who are eligible to receive preoperative chemotherapy.

DETAILED DESCRIPTION:
In this study, MRI will be used to determine the effects of pre-surgical chemotherapy on breast cancer. MRS looks at the chemical components of tissue. MRS may be helpful in understanding how pre-surgical chemotherapy works.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Blood (about 1 teaspoon) will be drawn for routine tests. Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test.

If you are found to be eligible to take part in this study, you will have 3 MRI with MRS scans on both breast including the affected breast. The scans will be performed before chemotherapy, 21 days (plus or minus 3 days) after you start chemotherapy (Day 1 = your first day of chemotherapy), and at the end of the chemotherapy/before surgery. If you have never had an MRI scan before, you will be given the opportunity to watch a 10-minute video to prepare you for the procedure.

You will have specialized MRI scans: MRS, DCE, and DW. The DCE is a Dynamic Contrast Enhanced MRI. DCE-MRI is used to create a 3-D image of the breast tumor, so that the small blood vessels can be seen. The Diffusion-Weighted (DW) MRI may possibly be used to study the structure of tumor cells based on the movement of water molecules in tumor tissue.

For this, you will lie still on your stomach with your breasts positioned within the openings of the detector. A contrast drug, which helps the MRI scanner to show the breast lesion, will be injected through a needle in your vein. The procedure will take about 1 hour.

The tissues removed during the surgery will be collected as part of this study. Small pieces of tissues will be stained with special stains to give more information about the tumor (such as invasiveness, blood vessel supply, number of positive lymph nodes, tissue changes). Multiple sections of the tissues will be stained to make sure that all tissue areas of interest will be able to be compared with MRI/MRS images. The tissues then will be photographed and x-rayed.

You will be considered off-study 6 months after surgery. If you are unable to have surgery, you will be considered off-study 6 months after the last MRI with MRS.

This is an investigational study. The MRI with MRS scans are FDA approved and commercially available. The first and third scans will be part of routine patient care. The second scan is not part of routine care. Up to 28 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed stage II A-B or III A-C breast cancers who are scheduled to start systemic chemotherapy.
2. Patients must have a histological diagnosis of invasive breast cancer.
3. Patients whose extent of disease is determined by physical examination and conventional imaging (mammography and sonography).
4. Patients should have not received any previous chemotherapy for their newly diagnosed Stage II A-B or III A-C breast cancer.
5. Patients must be age 18 or older.
6. ECOG performance status 0-2.
7. Patients with history of prior malignancies must be disease-free for at least 5 years prior of study entry.
8. Normal hematological function: WBC > 3000/ul, absolute neutrophil count > 1500/ul, platelets > 100,000/ul, and Hgb > 10 gms (transfusion to achieve Hgb > 10 gms is acceptable).
9. Serum total bilirubin < 1.5 mg/dl and SGPT < 1.5 X normal.
10. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policies of the hospital. The only acceptable consent form is the one attached at the end of this protocol.

Exclusion Criteria:

1. Patients who received previous chemotherapy for the newly diagnosed breast cancer.
2. Patients with no evidence of primary breast lesion (e.g., T0, Tx).
3. Patients who are unwilling to come back for regular assessments of response.
4. Patients with claustrophobia or obesity (exceeding the equipment weight limits).
5. Pregnant women, lactating women or sexually active women of childbearing potential who are not practicing adequate contraception.
6. Patients with myocardial infarction within 6 months of study entry; unstable angina pectoris; uncontrolled congestive heart failure; uncontrolled arrhythmias.
7. Patients with pacemakers or other metallic inserts that are not compatible with 3-T MR scanners.
8. Patients with bilateral breast disease, and recurrent newly diagnosed breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed stage II A-B or III A-C breast cancers who are scheduled to start systemic chemotherapy.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-10-25 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Individual Analyses between Quantitative MR Measures + Pathologic Outcome Measures | Before chemotherapy, 21 ± 3 days after the initiation of chemotherapy (day 1 = first day of chemotherapy), and at end of chemotherapy and prior to any surgery.
  Quantitative measures of tissue function obtained non-invasively by dynamic contrast enhanced (DCE) MRI, diffusion-weighted (DW) MRI, and proton MR spectroscopy (1H MRS) techniques to assess effects of pre-surgical chemotherapy in breast cancer patients eligible for preoperative chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Whitman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org